CLINICAL TRIAL: NCT05699447
Title: A New Risk Score for Predicting 1-year Mortality in Older r Maintenance Hemodialysis Patients.A Cohort Study in Beijing.
Brief Title: A New Risk Score for Predicting 1-year Mortality in Older r Maintenance Hemodialysis Patients.
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wenhu Liu, professor, Beijing Friendship Hospital
Other Study IDs: 2022-P2-385-01
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Maintenance Hemodialysis; Older Patient
Keywords: Older patients; maintenance hemodialysis; mortality; risk prediction score.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective observational cohort study is to analysis the 1-year mortality in older patients undergoing maintenance hemodialysis. The main question it aims to answer is to explore the risk factors affecting the mortality of older patients undergoing maintenance hemodialysis and establish a risk prediction score.

Data of older patients (age ≥65 years old) undergoing maintenance hemodialysis were collected from 2012-1-December 31, 2014, with data from Beijing Blood Purification Quality Control and Improvement Center (BJHDQCIC). Logistic regression model was used to evaluate the 1-year mortality and the influence of predictive factors. Internal validation of the model was performed using the bootstrap 1000 repeat sampling method. Area under receiver operating characteristic curve (AUC) was used to evaluate the predictive ability of the model.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years.
* More than 6-month history of hemodialysis,the frequency is 3 times a week, and the dialysis time is 4 hours each.
* The dialysate Ca concentration was 1.5 mmol/L and the bicarbonate level was 32 -- 35 mmol/L.

Exclusion Criteria:

* Lack of demographic information, clinical history, or relevant laboratory values (including pre-dialysis serum calcium, phosphorus, iPTH, haemoglobin, albumin, creatinine, total cholesterol, and Kt/v for urea).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Data of older patients (age ≥65 years old) undergoing maintenance hemodialysis were collected from 2012-1-December 31, 2014, with data from Beijing Blood Purification Quality Control and Improvement Center (BJHDQCIC).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
the 1-year mortality in older patients undergoing maintenance hemodialysis | Data of older patients (age ≥65 years old) undergoing maintenance hemodialysis were collected from 2012-1-December 31, 2014, with data from Beijing Blood Purification Quality Control and Improvement Center (BJHDQCIC).